CLINICAL TRIAL: NCT01255033
Title: Evaluation of the Continuous Measurement of Tissular (StO2) and Cerebral (ScO2) Oxygenation During Lung Surgery and During the 6 First Postoperative Hours (Prospective Monocentric Study).
Brief Title: Oxygen Peripheral Saturations and Lung Surgery
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/09
Record Dates: First submitted 2010-12-05; First posted 2010-12-07 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Surgical Procedures; Recovery Period
Keywords: perioperative surgery; regional oxygenation; hypoxemia; brain hypoxemia; spectroscopy, near-infrared
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulmonary surgical patients: Patients submitted for scheduled lung surgery requiring one-lung ventilation
  Interventions: Device: Monitoring of tissular oxygenation

INTERVENTIONS:
Device: Monitoring of tissular oxygenation — Equanox: cerebral oxygenation by spectroscopy, near-infrared through forehead and noninvasive devices
  Inspectra: tissular oxygenation by spectroscopy, near-infrared through thenar and noninvasive device

SUMMARY:
The purpose of this study is to compare the ability of two peripheral and non invasive devices to detect hypoxic events during one-lung ventilation and during the early postoperative period. One device measures regional cerebral oxygenation and the other muscular oxygenation. These two devices are compared to non invasive arterial saturation (SpO2), which is the gold standard.

DETAILED DESCRIPTION:
Lung surgery is often complicated by hypoxic evants :

* during one-lung ventilation which leads to changes about ratio in ventilated and perfused lung areas. This blood flow redistribution promotes shunt with a decreased arterial oxygenation and possible hypoxemia.
* during the postoperative period.

Common measure of arterial saturation through SpO2 may miss a great number of hypoxic events with regional impact because a significant decrease in SpO2 occurs for an arterial pressure in oxygen below 60 mmHg. Currently, cerebral and somatic saturation can be monitored non-invasively and continuously via optical sensors applied to the right and left forehead and to the thenar eminence. These devices may help clinicians in the detection of such hypoxemic events.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled lung surgery requiring one-lung ventilation
* informed consent

Exclusion Criteria:

* Pregnant woman
* Neurologic or psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted for scheduled lung surgery requiring one-lung ventilation
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Desaturation during surgery and early postoperative recovery whatever the device. | 6 hours postoperative
  Number of episodes

SECONDARY OUTCOMES:
Chronology between devices in case of desaturation | 6 hours post operative
Quality of signal | 6 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, Study Chair — Hôpital Foch
Locations (1):
- Hôpital Foch, Suresnes, France, France

REFERENCES:
- [Background] Manfredini F, Malagoni AM, Felisatti M, Mandini S, Mascoli F, Manfredini R, Basaglia N, Zamboni P. A dynamic objective evaluation of peripheral arterial disease by near-infrared spectroscopy. Eur J Vasc Endovasc Surg. 2009 Oct;38(4):441-8. doi: 10.1016/j.ejvs.2009.06.011. Epub 2009 Jul 21. PMID 19625198
- [Background] Mesquida J, Masip J, Gili G, Artigas A, Baigorri F. Thenar oxygen saturation measured by near infrared spectroscopy as a noninvasive predictor of low central venous oxygen saturation in septic patients. Intensive Care Med. 2009 Jun;35(6):1106-9. doi: 10.1007/s00134-009-1410-y. Epub 2009 Jan 29. PMID 19183952
- [Result] Kazan R, Bracco D, Hemmerling TM. Reduced cerebral oxygen saturation measured by absolute cerebral oximetry during thoracic surgery correlates with postoperative complications. Br J Anaesth. 2009 Dec;103(6):811-6. doi: 10.1093/bja/aep309. PMID 19918024
- [Result] Hemmerling TM, Kazan R, Bracco D. Inter-hemispheric cerebral oxygen saturation differences during thoracic surgery in lateral head positioning. Br J Anaesth. 2009 Jan;102(1):141-2. doi: 10.1093/bja/aen336. No abstract available. PMID 19059925